CLINICAL TRIAL: NCT06059053
Title: Outcome of the Semibranch in Pararenal and Thoracoabdominal Aortic Pathologies. A Prospective, Multicentre Registry.
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Alexander Oberhuber, Univ.-Prof. Dr. med. Alexander Oberhuber, University Hospital Muenster
Other Study IDs: Semibranch_Reg
Record Dates: First submitted 2023-09-14; First posted 2023-09-28 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Aortic Aneurysm; Endovascular Aortic Repair; Stent-Graft Endoleak
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Semibranch CMD branched aortic stentgraft — bEVAR with a custom made abdominal aortic multibranch, which incorporates the semibranch design

SUMMARY:
The goal of this registry is to evaluate the semibranch in branched endovascular aortic repair, which is a new tool in endovascular branched aortic repair.

DETAILED DESCRIPTION:
The main question it aims to answer are:

* Patency of the semibranch
* Feasibility of the technique regarding cannulation and stentgrafting

The participants will treated with the custom made semibranch device and enrolled in the registry if they consent. No change in treatment will be made when enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Presence of pararenal or thoracoabdominal aortic pathology
* Treatment planned a semibranch device branch from Artivion
* Availability of the patients during the follow up period
* Informing patients about the study and providing written informed consent

Exclusion Criteria:

* Women of childbearing age
* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pararenal or thoracoabdominal aortic pathology, who are treated with a endovascular semibranch stentgraft.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from target vessel instability | 30 days after intervention
  primary patency and freedom from stenosis fo the semibranch
Mortality | 30 days after intervention
  overall mortality rate during 30 days after intervention
technical success | During intervention
  Feasibility in terms of cannulation and stentgrafting of the semibranches

SECONDARY OUTCOMES:
Morbidity | During follow up period (up to 3 years)
  Access site, bowel ischemia, kidney failure, paraplegia
freedom Endoleak Type I and III | During follow up period (up to 3 years)
  absence of endoleaks arising from the semibranch
Long term mortality | During follow up period (up to 3 years)
  overall mortality up to 3 years
Branch patency | During follow up period (up to 3 years)
  primary patency of all branches

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Oberhuber, MD,PhD, Study Chair — Department of Vascular and Endovascular Surgery University Hospital Münster; Alexander Oberhuber, MD,PhD, Principal Investigator — Department of Vascular and Endovascular Surgery University Hospital Münster
Locations (1):
- Muenster University Hospital, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided